CLINICAL TRIAL: NCT07129551
Title: Navigation, Outcomes and Quality-of-life in Prostate Cancer Patients Undergoing PSMA-targeted Surgery
Acronym: NICE-PSMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Martini-Klinik am UKE GmbH (Other)
Responsible Party: Principal Investigator, Anke Renter, Studycoordinator, Martini-Klinik am UKE GmbH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-PS-02
Record Dates: First submitted 2025-08-05; First posted 2025-08-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer (Adenocarcinoma)
Keywords: PSMA; targeted surgery; radioguided surgery; 3D model navigation
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preop virtual 3D model (Experimental): Cohort A: Radical prostatectomy with PSMA-targeted lymph node dissection (separate specimen) and bilateral extended pelvic lymph node dissection with additional use of a virtual 3D-model (of preoperative PSMA-PET examination) prior to surgery and postoperatively; Cohort B: Salvage lymph node dissection with PSMA-targeted lymph node dissection (separate specimen) and at least ipsilateral pelvic template lymph node dissection with additional use of a virtual 3D-model (of preoperative PSMA-PET examination) prior to surgery and postoperatively
  Interventions: Procedure: preop virtual 3D model
- Control Intervention (Active Comparator): Cohort A: Radical prostatectomy with PSMA-targeted lymph node dissection (separate specimen) and bilateral extended pelvic lymph node dissection with use of standard PSMA-PET examination prior to surgery; only postoperatively a virtual 3D-model (of preoperative PSMA-PET examination) will be evaluated; Cohort B: Salvage lymph node dissection with PSMA-targeted lymph node dissection (separate specimen) and at least ipsilateral pelvic template lymph node dissection with use of standard PSMA-PET examination prior to surgery; only postoperatively a virtual 3D-model (of preoperative PSMA-PET examination) will be evaluated
  Interventions: Procedure: postop 3D model

INTERVENTIONS:
Procedure: preop virtual 3D model — Cohort A: Radical prostatectomy with PSMA-targeted lymph node dissection (separate specimen) and bilateral extended pelvic lymph node dissection with additional use of a virtual 3D-model (of preoperative PSMA-PET examination) prior to surgery and postoperatively; Cohort B: Salvage lymph node dissection with PSMA-targeted lymph node dissection (separate specimen) and at least ipsilateral pelvic template lymph node dissection with additional use of a virtual 3D-model (of preoperative PSMA-PET examination) prior to surgery and postoperatively
  Arms: preop virtual 3D model
Procedure: postop 3D model — Cohort A: Radical prostatectomy with PSMA-targeted lymph node dissection (separate specimen) and bilateral extended pelvic lymph node dissection with use of standard PSMA-PET examination prior to surgery; only postoperatively a virtual 3D-model (of preoperative PSMA-PET examination) will be evaluated; Cohort B: Salvage lymph node dissection with PSMA-targeted lymph node dissection (separate specimen) and at least ipsilateral pelvic template lymph node dissection with use of standard PSMA-PET examination prior to surgery; only postoperatively a virtual 3D-model (of preoperative PSMA-PET examination) will be evaluated
  Arms: Control Intervention

SUMMARY:
As part of a feasibility study, it's planned to use a 3D virtual mixed reality model with prostate cancer patients who show signs of lymph node metastasis and are scheduled for surgery. The model is based on PSMA PET imaging performed prior to surgery and will be evaluated by surgeons, the surgical team, and patients as part of the consultation process. First, the researcher investigates whether the removal of lymph node metastases has improved compared to the data in the literature . In addition, the study examines how the 3D model influences the movement of surgical instruments and the efficiency of surgical removal of lymph node metastases. To this end, the analyzed recorded video and position data of the instruments used during procedures performed with a surgical robot. It's also an aim to develop two methods-using landmarks and visual position tracking-for more targeted navigation during surgery. Additionally, short-term results examine, such as PSA response rates, as an indication of successful lymph node metastasis removal and patient quality of life.

DETAILED DESCRIPTION:
In this prospective feasibility study, it's planned to use a 3D virtual mixed reality model based on the preoperative PSMA PET. The model will be evaluated as an educational tool for patients and surgeons in cases of primary high-risk prostate cancer and prostate cancer recurrence with PSMA PET-positive lymph node metastasis. In general, the detection rate of PSMA-guided surgical procedures will investigate with the histological result as the reference. Furthermore, the influence of 3D visualization on the movement of surgical instruments and the efficiency of targeted resection is analyzed the help of image data from two cameras and the position data of the instruments during robot-assisted procedures. Additionally, will the investigators develop and examine two navigation methods (landmark-based registration and visual tracking) in a retrospective approach that use the preoperative PSMA PET and the image and instrument position data captured during robotic procedures. The short-term oncological outcomes (PSA response rates) will examine as an indicator of the successful removal of macroscopic PSMA-PET-positive lesions and the quality of life (QoL) of patients.

ELIGIBILITY:
Inclusion Criteria:

Cohort A:

* Patients with hormone-sensitive prostate cancer scheduled for radical prostatectomy with pelvic lymph node dissection
* <3 PSMA-PET-avid lymph node metastases (PSMA expression score >2) in the pelvis.

Cohort B:

* Patients with hormone-sensitive recurrent prostate cancer after radical prostatectomy with planned pelvic salvage lymph node dissection
* <3 PSMA-PET-avid lymph node metastases (PSMA expression score >2) in the pelvis
* PSA value <2ng/ml.

Exclusion Criteria:

* Estimated life expectancy <10 years
* contraindication for surgical intervention
* androgen deprivation therapy (ADT) within the last 3 months

Ages: 18 Years to 78 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 102 (Estimated)
Dates: Start 2026-01-21 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the detection rate of lymph node metastases using PSMA-targeted surgery with or without a virtual 3D model (the preoperative PSMA PET scan). | two weeks post surgery
  The 3D model is used for surgical guidance during open/robotic primary prostatectomy with pelvic lymph node dissection (Cohort A) or open/robotic salvage lymph node dissection (SLND) for recurrent prostate cancer (Cohort B). The postoperative histology of the specifically dissected tissue serves as a reference.

SECONDARY OUTCOMES:
Feasibility and accuracy of preoperative virtual 3D modeling for patient consultation and surgical planning (determined by pre- and postoperative standardized User Experience Questionnaire (UEQ) and Mixed reality Questionnaire). | six months after surgery
  Here, UEQ and Mixed realty Questionaires are evaluated. Here, no comparisons are made between randomized groups as the questionaires are only answered after presentation of the model. This endpoint is only evaluated in a descriptive manner reporting the values of each question within the questionaires (on a scale from 1-7 for the UEQ and 1-5 for the Mixed reality Questionaire)
Retrospective analysis of vision-based and robotic tracking methods for target detection and retrospective analysis of the efficiency of PSMA-targeted dissection based on instrument tracking information (in robotic surgery) | six months after surgery
  Here, only for robotic procedures intraoperative tracking of the instruments will be recorded via the simultaneous recording of the two camera lenses of the robotic camera system as well as by the provided access of instrument movements. The recordings as well as the movement towards the PSMA PET positive lesion intraoperatively will be evaluated in the whole population and, if feasible, also for the patient cohorts with or without prior 3D model visualization
Diagnostic accuracy of PSMA-PET-CT for detection of lymph node metastases during open/robotic primary prostatectomy with pelvic lymph node dissection (Cohort A) or open/robotic salvage lymph node dissection (SLND) for recurrent prostate cancer (Cohort B) | six months after surgery
  Here, as secondary outcome measurement the findings of properative PSMA-PET/CT will be compared with post-operative histology on a patient-side basis and at region-level (external iliac, obturator, internal iliac, common iliac, other locations) providing then results for true positive, false positive, true negative and false negative evaluations
Short-term oncologic outcomes (complete biochemical response (cBR), defined as a PSA level <0.2 ng/mL at 8-12 weeks (Cohort A) or 4-6 weeks (Cohort B)). | three months after surgery
  Here, percentages (0-100%) of complete biochemical response at the predefined timepoints will be evaluated in between both cohorts, comparing the randomized groups
Quality of life (SF-12, EPIC-26), morbidity (intra- and postoperative complications within 6 months according to the Clavien-Dindo classification) and satisfaction (Decision Regret Scale) after surgery | six months after surgery
  Here, standardized questionaires (SF-12, EPIC-26; mostly 5-scale evaluations) will be evaluated. Morbidity will be recorded according to Clavien-Dindo (CTC 1-5). Decision regret is evaluated according to the DRS (5-scale evaluations). Here, first the whole cohorts will be reported and then comparisons within the randomized groups in cohort A and B are made.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Martini-Klinik, Hamburg, Hamburg
  - Anke Renter, Hamburg, Hamburg

IPD SHARING:
Plan to Share IPD: No